CLINICAL TRIAL: NCT03234283
Title: Video-laryngoscopic Visualization of the Intubation Pathway With the "IRRIS"-Device. A Clinical Safety and Proof of Concept Study
Brief Title: Visualization of the Intubation Pathway With the "IRRIS"-Device
Acronym: IRRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-01657
Record Dates: First submitted 2017-05-18; First posted 2017-07-31 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Difficult Intubation
Keywords: Intubation

STUDY DESIGN:
Intervention Model Description: A prospective, open label, non-randomized, safety and feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study intervention group (Experimental): All participants will be intubated with a video-laryngiscope by guiding the tracheal tube according to the highlighted Larynx on the Video Screen.
  Interventions: Device: IRRIS InfraRed - Red Intubation System

INTERVENTIONS:
Device: IRRIS InfraRed - Red Intubation System — IRRIS will be attached to the patient's neck skin just beneath the laryngeal prominence. Tracheal intubation will be performed by using a video-laryngoscope in a standardized Fashion and by guiding the tracheal tube into the Larynx by following the visual Signal on the Screen that is caused by IRRIS. The handling of IRRIS and the Performance of tracheal Intubation will be recorded. Patients will be monitored for safety parameters and possible adverse events during the study until recovered and released from the postoperative care unit.

SUMMARY:
A prospective, open label, non-randomized, single centre safety and feasibility study. Patients with no expected airway difficulties scheduled for elective surgery including tracheal intubation and general anesthesia procedures will be enrolled into the study. Following standard induction of anesthesia, the IRRIS will be attached to the patient's neck skin just beneath the laryngeal prominence (Adam's apple) and the intubation will be performed by using a video-laryngoscope in a standardized fashion. The IRRIS device emits a light that penetrates through the skin into the airway and that is visible on the video-laryngoscope display. This light highlights the right pathway for the tracheal tube and facilitates the visual recognition and identification of the laryngeal inlet. In case of problems identified during the induction period such as an unexpected difficult intubation situation and the IRRIS does not provide the expected facilitation of intubation, the local "unexpected difficult airway" protocol goes into effect.

DETAILED DESCRIPTION:
The IRRIS (InfraRed - Red Intubation System) is an external disposable light source in a patch that is intended for single use while it is placed externally on the patient's neck before tracheal intubation for the duration of tracheal intubation. The device transmits near-infrared light through the skin towards the trachea. During laryngoscopy, the emitted light becomes visible only from the trachea and not from the oesophagus. Video assisted devices which already are in the market known as video-laryngoscopes and fiberoptic bronchoscopes are capable of detecting and visualizing the emitted light so that the anaesthesiologist who is performing the intubation is aided to direct and insert the endotracheal tube into the trachea by following the light on the screen of his video-assisted endoscope. The objective of this study is to assess the safety, and performance of IRRIS in patients who undergo tracheal intubation in terms of skin integrity, duration of intubation, number of attempts, success of intubation and usability aspects in terms of subjective physician grading of the IRRIS.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients scheduled for elective surgery requiring general anesthesia and tracheal intubation.
2. Patient age: adult (>18 years old)
3. Mallampati scores 1 to 3.
4. ASA Physical Status Classification System 1-3
5. Ability to understand the requirements of the study, willingness to comply with its instructions and schedules, and agreement to the informed consent

Exclusion Criteria:

1. Emergency cases
2. Expected airway difficulties as defined during the pre-anaesthesia visit
3. Necessity for an alternative airway management approach other than by using a video-laryngoscope
4. Rapid sequence induction
5. Skin disorders and skin light sensitivity (SLE, lupus, Porphyria, Dermatomyositis, Pemphigus, Pellagra etc.)
6. Known history of any significant medical disorder, which in the investigator's judgment contraindicates the patient's participation
7. Impaired head and neck mobility
8. Scars or skin injuries at the neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Safety 1: Absence of skin lesions | 15 minutes after end of anesthesia
  skin lesions, irritations after removal of the patch at the end of anesthesia (yes / no)
Safety 2: Severity of skin lesions | 15 minutes after end of anesthesia
  skin lesions, irritations after removal of the patch at the end of anesthesia (mild/moderate/severe)

SECONDARY OUTCOMES:
Proof of Concept 2: Intubation success | 5 minutes after start of intubation
  Successful video-laryngoscopic tracheal intubation
Proof of Concept 3: Intubation success | 5 minutes after start of intubation
  Duration of intubation (time in seconds from inserting the video laryngoscope till tracheal tube cuff inflation)
Proof of Concept 4: Intubation success | 5 minutes after start of intubation
  Number of video laryngoscopy attempts till successful tracheal tube placement (number of video laryngoscope insertions during an intubation process that are related to the IRRIS operation)
Proof of Concept 5: Ease of use of IRRIS | 5 minutes after start of intubation
  Subjective degree of difficulty of the entire intubation process according a Verbal Rating Scale (VRS) assessed by the intubation person (values from 1 = very easy to 10 = extremely difficult)
Proof of Concept 7: Ease of use of IRRIS | 5 minutes after start of intubation
  Subjective degree of helpfulness of the visual aid by the device: according a Verbal Rating Scale (VRS) assessed by the intubation person (values from 1 = not helpful at all to 10 = very helpful)
Proof of Concept 8: Intubation success | 5 minutes after start of intubation
  Failures: necessity of alternative airway securing or abort of tracheal intubation if initial attempt(s) with IRRIS failed. (yes / no and number and choice of alternative techniques)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Biro, MD, Principal Investigator — University Hospital Zurich, Institue of Anesthesiology
Locations (1):
- University Hospital Zurich, Institue of Anesthesiology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goto Y, Goto T, Hagiwara Y, Tsugawa Y, Watase H, Okamoto H, Hasegawa K; Japanese Emergency Medicine Network Investigators. Techniques and outcomes of emergency airway management in Japan: An analysis of two multicentre prospective observational studies, 2010-2016. Resuscitation. 2017 May;114:14-20. doi: 10.1016/j.resuscitation.2017.02.009. Epub 2017 Feb 17. PMID 28219617
- [Result] Brown CA 3rd, Bair AE, Pallin DJ, Walls RM; NEAR III Investigators. Techniques, success, and adverse events of emergency department adult intubations. Ann Emerg Med. 2015 Apr;65(4):363-370.e1. doi: 10.1016/j.annemergmed.2014.10.036. Epub 2014 Dec 20. PMID 25533140
- [Result] Howard-Quijano KJ, Huang YM, Matevosian R, Kaplan MB, Steadman RH. Video-assisted instruction improves the success rate for tracheal intubation by novices. Br J Anaesth. 2008 Oct;101(4):568-72. doi: 10.1093/bja/aen211. Epub 2008 Aug 1. PMID 18676418
- [Result] Song Y, Oh J, Chee Y, Lim T, Kang H, Cho Y. A novel method to position an endotracheal tube at the correct depth using an infrared sensor stylet. Can J Anaesth. 2013 May;60(5):444-9. doi: 10.1007/s12630-013-9898-6. Epub 2013 Feb 1. PMID 23370979
- [Result] El-Sayed IH, Ho JE, Eisele DW. External light guidance for percutaneous dilatational tracheotomy. Head Neck. 2011 Aug;33(8):1206-9. doi: 10.1002/hed.21610. Epub 2011 Mar 16. PMID 21413098
- [Result] Kaplan MB, Ward D, Hagberg CA, Berci G, Hagiike M. Seeing is believing: the importance of video laryngoscopy in teaching and in managing the difficult airway. Surg Endosc. 2006 Apr;20 Suppl 2:S479-83. doi: 10.1007/s00464-006-0038-z. Epub 2006 Mar 16. PMID 16544062